CLINICAL TRIAL: NCT02448875
Title: Randomized, Prospective Clinical Evaluation of the Safety and Effectiveness of Visco-Assisted CyPass® Implantation in Patients With Open Angle Glaucoma
Brief Title: Clinical Evaluation of Visco-Assisted CyPass® Micro-Stent Implantation in Patients With Open Angle Glaucoma
Acronym: ViscoPass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMI-13-01; GLD122-P001 (Other: Alcon)
Record Dates: First submitted 2015-05-12; First posted 2015-05-20 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- CyPass (Active Comparator): CyPass Micro-Stent without adjunct viscoelastic implanted in the study eye
  Interventions: Device: CyPass Micro-Stent
- CyPass30 (Experimental): CyPass Micro-Stent implantation followed by targeted delivery of 30 μl ophthalmic viscoelastic
  Interventions: Device: CyPass Micro-Stent; Device: Viscoelastic
- CyPass60 (Experimental): CyPass Micro-Stent implantation followed by targeted delivery of 60 μl ophthalmic viscoelastic
  Interventions: Device: CyPass Micro-Stent; Device: Viscoelastic

INTERVENTIONS:
Device: CyPass Micro-Stent — Small tube with a through-lumen designed to redirect aqueous fluid from the front to the back of the eye in order to reduce intraocular pressure. Designed to be permanently implanted in the eye.
  Other Names: Model 2FX
Device: Viscoelastic — Healon 5 ophthalmic viscoelastic used to increase the size of the aqueous drainage area created by the CyPass Micro-Stent
  Arms: CyPass30; CyPass60

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the use of visco-assisted CyPass® Micro-Stent implantation for the lowering of intraocular pressure (IOP) in subjects who have open angle glaucoma (OAG).

DETAILED DESCRIPTION:
The study was conducted in 2 phases. Only one eye per subject was treated for each independent phase.

Dose Selection Phase (Cohort 1): Subjects were randomized in a 1:1:1 ratio and implanted with either a CyPass Micro-Stent with targeted delivery of 30 microliters (μl) ophthalmic 5 viscoelastic, a CyPass Micro-Stent with targeted delivery of 60 μl of ophthalmic viscoelastic, or a CyPass Micro-Stent without adjunct viscoelastic in the study eye.

Expansion Phase (Cohort 2): Subjects were randomized in a 1:1 ratio and implanted with either the CyPass Micro-Stent without adjunct viscoelastic or the CyPass Micro-Stent with 60 μl of ophthalmic viscoelastic (based on Dose Selection results). Subjects were randomized to treatment on the day of their surgical procedure. A total of 9 scheduled visits were planned including Screening (Day -45 to -2), Baseline (Day -15 to -1), Surgery (Day 0), 1 Day (Day 1), 1 Week (Day 5-9), 1 Month (Day 21-35), 3 Month (Day 70-98), 6 Month (Day 150-210), and 12 Month (Day 330-420) visits. The total expected duration of participation for each subject was up to 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma;
* Unmedicated IOP between 21 - 36 mmHg, inclusive;
* Normal angle anatomy at site of intended CyPass Micro-Stent implantation.

Exclusion Criteria:

* Advanced glaucoma;
* Prior incisional glaucoma surgery;
* Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma;
* Clinically significant ocular pathology other than glaucoma.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (6):
- Germany (3):
  - Transcend Medical Investigative Site, Lübeck
  - Transcend Medical Investigative Site, Mainz
  - Transcend Medical Investigative Site, Neubrandenburg
- Transcend Medical Investigative Site, Panama City, Panama
- Transcend Medical Investigative Site, Warsaw, Poland
- Transcend Medical Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study centers located in Germany (3), Poland (1), Spain (1), and Panama (1).
Pre-assignment Details: Of the 192 enrolled, 49 subjects were exited prior to randomization. In addition, one randomized subject discontinued prior to treatment. This reporting group includes all treated subjects, Dose Selection Phase and Expansion Phase (142 subjects).
Period: Overall Study
Arm/Group | CyPass | CyPass30 | CyPass60
Started (Includes dose selection phase and expansion phase) | 60 | 21 | 61
Completed Dose Selection Phase | 20 | 21 | 20
Full Analysis Set | 60 | 21 | 61
Safety Analysis Set | 60 | 21 | 61
Completed (Completed expansion phase) | 53 | 20 | 60
Not Completed | 7 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Investigator Decision | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | CyPass | CyPass30 | CyPass60 | Total
Number analyzed (Participants) | 60 | 21 | 61 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.87) | 68.7 (9.68) | 65.4 (11.17) | 65.9 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 11 | 29 | 77
  Male | 23 | 10 | 32 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 5 | 36 | 73
  Black or African American | 10 | 5 | 2 | 17
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 18 | 11 | 23 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥ 20% Decrease From Baseline to 12 Months Postoperative in IOP Without Use of Ocular Hypotensive Medication
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) contributed to the analysis. No formal statistical hypothesis testing was planned for the study.
Time Frame: Baseline (Day -1), Month 12 PostOperative
Population: Full Analysis Set with data available
Measure: Number; unit: percentage of subjects
Arm/Group | CyPass | CyPass30 | CyPass60
Number analyzed (Participants) | 46 | 12 | 49
percentage of subjects | 63.0 | 83.3 | 73.5

2. Secondary Outcome: Percentage of Subjects With Device-related Ocular Adverse Events
Description: A device related adverse event (AE) was any AE that was considered to be possibly, probably, or definitely related to the device in the opinion of the investigator. Reported categorically as intraoperative (start date on the date of surgery) and postoperative (start date after surgery). One eye (study eye) contributed to the analysis. No formal statistical hypothesis testing was planned for the study.
Time Frame: Up to Month 12 PostOperative
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | CyPass | CyPass30 | CyPass60
Number analyzed (Participants) | 60 | 21 | 61
percentage of subjects
  Intraoperative | 1.7 | 4.8 | 4.9
  Postoperative | 58.3 | 71.4 | 63.9

3. Secondary Outcome: Mean Change From Baseline to 12 Months Postoperative in Medicated IOP
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A higher negative change indicates improvement. One eye (study eye) contributed to the analysis. No formal statistical hypothesis testing was planned for the study.
Time Frame: Baseline (Day -1), Month 12 PostOperative
Population: Full Analysis Set with data available
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | CyPass | CyPass30 | CyPass60
Number analyzed (Participants) | 60 | 21 | 60
millimeters of mercury (mmHg)
  Baseline | 21.08 (5.004) | 22.17 (6.683) | 21.71 (5.279)
  Change from Baseline @ Month 12: number analyzed (Participants) | 56 | 21 | 60
  Change from Baseline @ Month 12 | -4.29 (5.360) | -4.00 (6.736) | -4.81 (6.406)

4. Secondary Outcome: Percentage of Eyes Using Ocular Hypotensive Medication at 12 Months
Description: The use of ocular hypotensive medications was assessed in subjects with at least one IOP-lowering medication at 12 Months. One eye (study eye) contributed to the analysis. No formal statistical hypothesis testing was planned for the study.
Time Frame: Month 12 PostOperative
Population: Full Analysis Set with data available
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | CyPass | CyPass30 | CyPass60
Number analyzed (Participants) | 56 | 21 | 61
Number analyzed (Eyes) | 56 | 21 | 61
percentage of eyes | 37.5 | 42.9 | 36.1

5. Secondary Outcome: Mean Change From Screening to 12 Months Postoperative in Number of Topical IOP-lowering Medications Used
Description: The number of IOP lowering medications in subjects at 12 months was compared to medicated baseline. A higher negative change indicates improvement. One eye (study eye) contributed to the analysis. No formal statistical hypothesis testing was planned for the study.
Time Frame: Screening (Day -2), Month 12 PostOperative
Population: Full Analysis Set with data available
Measure: Mean (Standard Deviation); unit: IOP-lowering medications
Arm/Group | CyPass | CyPass30 | CyPass60
Number analyzed (Participants) | 56 | 21 | 61
IOP-lowering medications | -0.8 (1.38) | -0.3 (1.74) | -0.8 (1.47)

ADVERSE EVENTS:
Time Frame: Surgery through study completion, an average of 12 months.
Description: Safety was assessed at each study visit. The Safety Analysis Set was used for this analysis.
Groups:
- CyPass Ocular; CyPass Nonocular: Subjects with CyPass Micro-Stent implantation
- CyPass30 Ocular; CyPass30 Nonocular: Subjects with CyPass Micro-Stent implantation followed by targeted delivery of 30 μl ophthalmic viscoelastic
- CyPass60 Ocular; CyPass60 Nonocular: Subjects with CyPass Micro-Stent implantation followed by targeted delivery of 60 μl ophthalmic viscoelastic
Arm/Group | CyPass Ocular | CyPass Nonocular | CyPass30 Ocular | CyPass30 Nonocular | CyPass60 Ocular | CyPass60 Nonocular
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/21 | 0/21 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 6/60 | 4/60 | 1/21 | 0/21 | 7/61 | 2/61
Other Adverse Events (participants affected / at risk) | 38/60 | 0/60 | 13/21 | 0/21 | 37/61 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Ocular (N=60) | CyPass Nonocular (N=60) | CyPass30 Ocular (N=21) | CyPass30 Nonocular (N=21) | CyPass60 Ocular (N=61) | CyPass60 Nonocular (N=61)
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotony of eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0 | 0 | 3 | 0
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Intraocular pressure fluctuation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 4 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Ocular (N=60) | CyPass Nonocular (N=60) | CyPass30 Ocular (N=21) | CyPass30 Nonocular (N=21) | CyPass60 Ocular (N=61) | CyPass60 Nonocular (N=61)
Cataract (Eye disorders) | 13 | 0 | 3 | 0 | 14 | 0
Visual acuity reduced (Eye disorders) | 20 | 0 | 7 | 0 | 19 | 0
Intraocular pressure increased (Investigations) | 11 | 0 | 3 | 0 | 9 | 0
Device occlusion (Product Issues) | 12 | 0 | 8 | 0 | 18 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2014-10-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02448875/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT02448875/SAP_001.pdf